CLINICAL TRIAL: NCT00543920
Title: A Study of MK0777 in the Treatment of Outpatients With Generalized Anxiety Disorder (0777-020)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0777-020; 2007_633
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — 7-(1,1-dimethylethyl)-6-(2-ethyl-2H-1,2,4-triazol-3-ylmethoxy)-3-(2-fluorophenyl)-1,2,4-triazolo(4,3-b)pyridazine

INTERVENTIONS:
Drug: MK0777

SUMMARY:
The study will look at the effect of MK0777on reducing anxiety in subjects with general anxiety disorder.

This is an early phase trial and some specific protocol information is in progress and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of General Anxiety Order

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* History of severe drug reaction
* History of severe drug withdrawal symptoms such as seizures or delirium
* Disease of cardiovascular system
* Disease of the liver, kidneys, endocrine system, metabolic system or eyes
* History of seizures or seizure disorder
* History of drug or alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC